CLINICAL TRIAL: NCT05123846
Title: Medical Affairs Pharmaceutical Physician Work-related Quality of Life (MAPPWrQoL) Instrument Development and Patient Registry (MAPPWrQoLReg)
Status: Recruiting | Type: Observational
Sponsor: Medialis Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: KCL Asset 10 and 11
Record Dates: First submitted 2021-11-05; First posted 2021-11-17 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Quality of Life
Keywords: Quality of Life; Jandhyala Method; Medical Affairs; Occupational burnout; Stress; Anxiety
MeSH Terms: conditions — Burnout, Professional; Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Existing evidence has shown that medical affairs pharmaceutical physicians (MAPPs), are a core function within the pharmaceutical industry. Despite their expertise, there are ongoing concerns about recognition and respect for the MAPP's role within the pharmaceutical industry. Anecdotal evidence further suggests that this lack of recognition and respect for the valuable contribution of this specialised group of medical doctors may impact their quality of life, resulting in stress, anxiety, depression and occupational burnout. Hence, participants are likely to use NHS services as patients, when experiencing the physical, mental, and emotional issues associated with occupational burnout, an internationally recognised condition (ICD-11 code QD85) resulting from chronic occupational stress.

This observational study will recruit participants to contribute data to creating a MAPP work-related participant-reported outcome measure on the impact of work-related performance on quality of life (QoL). The created MAPP work-related participant-reported measure will be used longitudinally with study participants to measure their QoL monthly for 12 months. In total, up to 180 Medical Affairs Pharmaceutical Physicians are expected to be recruited to the study. The study will be conducted in two main phases, involving three online surveys.

DETAILED DESCRIPTION:
Phase One - the development of a MAPP work-related participant-reported quality of life (MAPPWrQoL) measure

The study will recruit between nine and 15 participants in this phase. Firstly, a novel method, the Jandhyala Method [16], will be used to elicit medical affairs pharmaceutical physicians' preferences for a QoL tool addressing work-related performance.

Below is the outline of activities to be completed during Phase One:

1. Awareness Round survey (first survey, hosted on Survey Monkey) - asking for areas of their life which the participants feel have been impacted by work-related performance, including details and examples of those impacts.
2. The research team will collate and code these responses and generate a list of statements based on the information provided by participants.
3. Consensus Round survey (second survey, hosted on Survey Monkey) - the list of statements will be sent to participants. Participants will be asked to rate their agreement or disagreement with the inclusion of these areas in a MAPP work-related QoL tool.
4. The research team will collate this information, group it into relevant domains and develop a weighting tool.
5. Weighting tool (online Microsoft excel template) - participants will be asked to assign a percentage value (as weights) to the individual items and domains for the finalised MAPP work-related QoL tool using an online excel spreadsheet template.
6. The research team will use this information to develop the finalised MAPP work-related QoL measure to be completed by participants and to develop the system to score this tool.

The research team expect the Awareness Round survey (first survey) to be completed within a month. Following this, two weeks will be allocated for the research team to analyse and finalise the survey to be used during the Consensus Round (second survey). The consensus Round survey will be open for two weeks, and participants will be prompted after one week if yet to complete the survey. We will send five reminder emails to the participants. The research team will have two weeks to complete the weighting tool, and participants will be given another two weeks to complete this. The research team will have an additional two weeks to finalise the MAPP work-related QoL at this stage. Thus, it is expected that Phase one activities will take up to 3 months to complete.

Phase two - the longitudinal completion of the quality of life tool by Medical Affairs Pharmaceutical Physicians each month for 12 months - observational patient study (MAPPWrQoLReg)

Following the MAPP work-related QoL tool development, the research team will recruit additional participants to complete the developed tool monthly for 12 months. The research team will aim to recruit a maximum of 165 study participants for this phase. Participants involved in Phase one will have the option to continue to Phase two. However, participation in Phase two is not a criterion for participation in Phase one. Recruitment will remain open for phase two for a minimum of one year and then reviewed, with another year following this to gain the full 12 months of data from participants.

The finalised MAPP work-related QoL measure will be hosted on a secure online system (Survey Monkey), and participants will be allocated an identification (ID) record number. Participants will be asked to complete this measure at monthly intervals for 12 months. Statistical methods for this phase will be finalised when the measure has been completed at the end of phase one by the Biostatistician Team at Medialis Ltd.

ELIGIBILITY:
Inclusion Criteria:

Phase one and Phase two: Participants will be eligible to take part in Phase One based on the following criteria:

* Qualification as a Medical Affairs Pharmaceutical Physician (qualified by medical degree).
* Previous or current work experience within a pharmaceutical company (industry-based).
* The participant can provide informed consent.
* The participant can read, write, and converse in English.
* The participant can comply with the study schedule.
* 18 years and above.

Exclusion Criteria:

* Non-industry based Medical Affairs Pharmaceutical Physicians
* Not able to comply with the study schedule
* Not able to read, write, and converse in English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participant are medical affairs pharmaceutical physicians, with pharmaceutical industry-based work experience.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2021-11-03 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Development and validation of MAPPWrQoL instrument. | 3 months.
  The design and creation of a work-related quality of life measure to be self-administered by medical affairs pharmaceutical physicians.
A prospective MAPPWrQoL patient registry. | 12 months
  Implementation of the developed MAPPWrQoL instrument as the core dataset in the associated patient registry (MAPPWrQoLReg).

CONTACTS AND LOCATIONS:
Overall Officials: Ravi Jandhyala, Principal Investigator — Medialis Ltd.
Locations (1):
- Medialis, Oxford, United Kingdom

REFERENCES:
- [Derived] Jandhyala R. Development, validation and implementation of the medical affairs pharmaceutical physician work-related quality of life instrument. Curr Med Res Opin. 2023 Dec;39(12):1567-1574. doi: 10.1080/03007995.2023.2174747. Epub 2023 Feb 8. PMID 36719367
- See also: Publication — https://www.frontiersin.org/articles/10.3389/fphar.2022.842431/full
- See also: Publication — https://link.springer.com/article/10.1007/s40290-021-00413-9